### STATISTICAL ANALYSIS PLAN

| Clinical Trial Protocol Identification No: | ITOLI-C19-02-I-00 |
|---|---|
| Title: | A Multi-Centric, Open label, Two Arm Randomized, Pivotal Phase2 Trial to Study the Efficacy and Safety of Itolizumab in COVID-19 Complications. |
| Trial Phase: | Pivotal Phase II |
| Name of the Drug: | Itolizumab (ALZUMAb <sup>TM</sup> ) |
| Clinical Trial Protocol Date and Version: | 3-June-2020/ Version 5.0 |
| Statistical Analysis Plan Date and Version: | 29-June-2020/ Final |
| Sponsor: | Biocon Biologics India Limited, Biocon House, Electronic City, Bengaluru – 560100, India |

#### CONFIDENTIALITY STATEMENT

The information in this document is a confidential communication of Biocon Biologics India Limited. Acceptance of this document constitutes an agreement by the recipient(s) that no unpublished information contained herein will be published or disclosed without prior written approval from Biocon Biologics India Limited.


#### **SIGNATURE PAGE**

#### Prepared by

Anjaiah Kalva Deputy Manager (CDMA Biostatistics) Biocon Biologics India Limited

Anjaiah Kalva

Digitally signed by Anjaiah Kalva Date: 2020.06.30 10:09:02 +05'30'

Signature

Date

### Reviewed & Approved by

Ashwani Marwah Sr. Manager (CDMA Biostatistics) Biocon Biologics India Limited

Ashwani Digitally signed by Ashwani Marwah Marwah

Date: 2020.06.30 10:14:57 +05'30'

Signature

Date

| Subramanian L<br>General Manager<br>Biocon Biologics | Sciences) | Subramanian | Loganathan | Digitally signed by Subramanian<br>Loganathan<br>Date: 2020.06.30 12:30:16 +05'30' |
|---|---|---|---|---|
| | _ | Signature | Date | |


# **Table of Contents**

| List | of ab | bbreviations | 6 |
|---|---|---|---|
| 1 | Purp | pose | 7 |
| 2 | Resp | sponsibility | 7 |
| 3 | Stud | dy Objectives | 7 |
| 3. | 1 | Trial Objectives | 7 |
| | 3.1. | .1 Primary Objectives | 7 |
| | 3.1.2 | 2 Secondary Objectives | 7 |
| 3. | 2 | Outcome Measures | 8 |
| | 3.2. | .1 Primary endpoint | 8 |
| | 3.2.2 | 2 Secondary endpoints | 8 |
| 4 | TRI | IAL DESIGN AND DESCRIPTION | 9 |
| 4. | 1 | Trial Design | 9 |
| 4. | 2 | Subject Selection | 9 |
| 4. | 3 | Inclusion Criteria | 9 |
| 4. | 4 | Exclusion Criteria | 9 |
| 4. | 5 | Sample Size, Treatment Assignment, Randomization | 10 |
| 5 | Prot | tocol Deviation | 10 |
| 6 | Gen | neral Aspects for Statistical Methods | 10 |
| 7 | Ana | alysis Population | 11 |
| 8 | Den | mography other baseline Characterstics | 11 |
| 9 | Effic | icacy Evaluation | 11 |
| 10 | О | Other Evaluations | 13 |
| 11 | In | nterim Study Report | 13 |
| 12 | K | Key Definitions | 13 |
| 13 | Pı | Programming Considerations, Listing of Tables, Figures & Format, Software detail | 14 |
| 14 | T | Tables and mock shells | 15 |
| 14.1 | .1 | Screening Failures | 15 |
| 14.1 | .2 | Disposition of Patients | 16 |
| 14.1 | .3 | Subject Disposition by Centre | 17 |
| 14.1 | .4 | Summary of Demographic Characterstics | 17 |
| 14.1 | .5 Su | ummary of Concomitant Medication by treatment group | 18 |
| 14.1 | .6 | Summary of Medical History | 18 |
| Conf | ident | · | |

| 14.1.7 Summa | ary of Vital Parameters and change from Baseline | 19 |
|---|---|---|
| 14.1.8 Summ | ary of Laboratory Test Results and Change from Baseline: Ho | ematology20 |
| 14.1.9 Summ | ary of Laboratory Test Results and Change from Baseline: Bi | iochemistry20 |
| 14.1.10 Hospital | ization | 22 |
| 14.1.11 Dura | ation of hospitalization and ICU stay | 23 |
| 14.1.12 Sum | nmary of Study Treatment: Itolizumab treatment details in Ar | m A24 |
| 14.1.13 Summar | y of BSC treatment details in both arms | 25 |
| 14.2 Primary out | tcome measures | 26 |
| 14.2.1 Primary C | Outcome Measures | 26 |
| 14.2.2 Proportion | n of patients needed intubation during the study | 26 |
| 14.2.3 Reduction | n in proportion of patients who need Non-invasive ventilation | 26 |
| 14.2.4 Reduction | n in proportion of patients who need NRBM | 27 |
| 14.2.5 Reduction | n in proportion of patients who need Face Mask | 27 |
| 14.2.6 Reduction | n in proportion of patients who need High Flow Nasal Oxyger | n28 |
| 14.2.7 One-mor | nth Mortality Rate | 28 |
| 14.2.8 Change | in inflammatory markers before and after dosing in Treatmen | t ARM A28 |
| 14.2.9 Survival s | status | 29 |
| 14.2.10 Summar | y of Oxygen and SOFA analysis | 29 |
| 14.2.11 Ordinal | Scale: No and Proportion of patient reduced by 1 or more poi | nts30 |
| 14.2.12 Improve | ment in respiratory rate | 30 |
| 14.3 Safety Anal | lysis | 31 |
| 14.3.1 Summary | of Subjects with TEAEs by treatment group | 31 |
| 14.3.2 Treatment | t Emergent Adverse Event (TEAE) by SOC and PT | 32 |
| 14.3.3 Treatment | t Emergent Adverse Event (TEAE) by severity | 33 |
| 14.3.4 Treatment | t Emergent Adverse Event (TEAE) related to study drug | 33 |
| 14.3.5 Treatment | t Emergent Adverse Event (TEAE) by Outcome | 33 |
| 15. Supplementa | ry Tables | 34 |
| 16. Listings | | 35 |
| Listing 16.1.1 St | ubjects Inclusion | 35 |
| Listing 16.1.2 Su | ubjects Exclusion | 35 |
| Listing 16.1.3 De | emographic data | 36 |
| Listing 16.1.4 M | edical History | 36 |
| Listing 16.1.5 Co | oncomitant Medication | 36 |

| Listing 16.1.6 Disposition of Subjects | 36 |
|----------------------------------------|----|
| Listing 16.1.7 Vital Parameters | 37 |
| Listing 16.1.8 Biomarker | 37 |
| Listing 16.1.9 Haematology | 37 |
| Listing 16.1.10 Biochemistry | 37 |
| Listing 16.1.13 Chest X Ray/CT Scan | 39 |
| Listing 16.1.14 Adverse Event (Part1) | 39 |
| Listing 16.1.15 Adverse Event (Part-2) | 39 |
| Listing 16.1.16 Hospitalization | 39 |
| Listing 16.1.17 Survival Status | 40 |
| Listing 16.1.18 SOFA Score | 40 |
| Listing 16.1.19 Ordinal Scale | 40 |
| Figure 1 Disposition by centres | 40 |
| Figure 2 PaO2/FiO2 ratio. | 40 |

#### List of abbreviations

| ADR | Adverse Drug Reaction |
|-----------|-------------------------------------------------------------|
| AE | Adverse event |
| ALT/SGPT/ | Alanine Transaminase / Serum Glutamic Pyruvic Transaminase/ |
| ALAT | Alanine Aminotransferase |
| ANC | Absolute Neutrophil Count |
| AP | Alkaline Phosphatase |
| AST / | Aspartate Transaminase/ Serum Glutamic Oxaloacetic |
| SGOT/ASAT | Transaminase/Aspartate Aminotransferase |
| ART | Adverse Reaction Terminology |
| CRO | Contract Research Organization |
| CSR | Clinical Study Report |
| CRP | (C-Reactive Protein) Level |
| ECG | Electrocardiogram |
| EOS | End of Study |
| ЕоТ | End of Trial |
| eCRF | Electronic case report form |
| FiO2 | Fraction of Inspired Oxygen |
| i.v. | intravenous(ly) |
| IMP | Investigational Medical Product |
| IRC | Independent Review Committee |
| IE | In evaluable |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PP | Per Protocol |
| PaO2 | Partial Pressure of Oxygen |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis System |
| SAP | Statistical Analysis Plan |
| UNK | Unknown |
| US | Ultrasound |
| V | Visit |
| Wk | Week |


#### 1 Purpose

The purpose of this statistical analysis plan (SAP) is to assess the efficacy and safety of Itolizumab administered in patients with COVID-19 complications in comparison with the Best of Care that will be included in the clinical study report. And this document is based on protocol version 5.0, 3rd June 2020. SAP will ensure that the data listings, summary tables and figures are complete; and the statistical methodologies used are appropriate to allow valid conclusions in line with the study's objectives. This document will be appended to the clinical study report (CSR). The statistical analyses will be performed in accordance with the ICH-E9 guidelines "Statistical Principles for Clinical Trials" and relevant guidelines from Central Drugs Standard Control organization (CDSCO). If circumstances arise during the study such that more appropriate analytic procedures become available, this statistical analysis plan (SAP) may be revised. Any revisions to the SAP (both alternative and additional methods) will be made prior to database lock and reasons for such revisions will be described in the final Clinical Study Report (CSR).

#### 2 Responsibility

Biocon Biologics India Limited/Designated CRO will be responsible for the conduct of statistical analyses, and the production and quality control of all tables, figures and listings).

#### 3 Study Objectives

Coronavirus disease 2019 (COVID-19) progresses to respiratory complications as consequence of the exaggerated immune response of the host, producing a pro-inflammatory cytokine storm syndrome (i.e.: IL-6, TNF) and cytopenia, with a high mortality rate. Emergency treatments aiming to reduce individual cytokines (IL-6 and IL-1) specifically [or indirectly (JAK inhibitors and CCR5 antagonists) have shown survival benefit in patients with hyperinflammation, without increased adverse events. However, not being sufficient to reduce the rising mortality by COVID-19 other interventions to immunomodulate the life-threatening hyperinflammation are urgently needed. Therefore, the proposal for use of an anti-CD6 monoclonal antibody (Itolizumab) for the treatment of the COVID-19 complications (cytokine storm syndrome).

#### 3.1 Trial Objectives

#### 3.1.1 Primary Objectives

To study the efficacy and safety of adding Itolizumab in patients with Moderate to Severe COVID-19 complications (Cytokine Release Syndrome).

#### 3.1.2 Secondary Objectives

To study the effect of immunomodulation by Itolizumab and its correlation to clinical improvement by evaluating biomarker data (IL6, TNF-a, IL17, IL1, Interferon -A etc.) before and after Itolizumab treatment


#### 3.2 Outcome Measures

#### 3.2.1 Primary endpoint

- 1. Proportion of patients with deterioration of lung function as measured by\*:
  - Stable SpO2 without increasing FiO2
  - Stable PaO2 without increasing FiO2
- 2. Reduction of endo-tracheal intubation rate, measured as rate of patients needing intubation\*
- 3. Reduction in proportion of patients who need\*
  - Non-invasive ventilation
  - Invasive mechanical ventilation
  - High flow nasal oxygen
- 4. Time of duration of mechanical ventilation or time to end of mechanical, measured as elapsed time from the start date of mechanical ventilation to the weaning date, for patients needing intubation\*
- 5. One-month mortality rate between the two arms\* [ Time Frame: up to 1 month ] 1-month mortality is defined as the ratio of patients who will live after 1month from study start out of those registered at baseline
- 6. Change in inflammatory markers like CRP (C-reactive protein) level, d-Dimer, ferritin etc. [Time Frame: Arm A; baseline, during treatment (Before every dose and 12 to 24 h after every dose) up to 1 month, Arm B: baseline, 12 to 24 h and approx. 7 and 14 days after randomization ]

#### 3.2.2 Secondary endpoints

- 1. Biomarkers (IL-6, TNF-a, IL1, IL17, etc...) [ Time Frame: Arm A; baseline, during treatment (Before every dose and 12 to 24 h post dose) up to 1 month, Arm B; baseline, 12 to 24 h and approx. 7 and 14 days after randomization ]
- 2. Lymphocyte count [ Time Frame: Arm A; baseline and before every dose up to 1 month, Arm B; baseline, approx. 7 and 14 days after randomization ] Lymphocyte count assessed by routinely used determination of blood count
- 3. PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio) [ Time Frame: Arm A; baseline, during treatment (Before every dose and 48 h post dose) up to 1 month, Arm B: baseline, 48 h and approx. 7 and 14 days after randomization] calculated from arterial blood gas analyses (values from 300 to 100)
- 4. Number of participants with treatment-related side effects as assessed by Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 [ Time Frame: during treatment and up to 30 days after the last treatment dose ]\* graded according to CTCAE citeria (v5.0)
- 5. Radiological response [ Time Frame: at baseline, after seven days and if clinically indicated (up to 1 month)]\* Thoracic CT scan or Chest XR
- 6. Duration of hospitalization [ Time Frame: from baseline up to patient's discharge (up to 1 month) ]\* Days of hospitalization and ICU


<sup>\*</sup> Applicable for both the arm

7. Remission of respiratory symptoms [ Time Frame: up to 1 month ]\* time to independence from non-invasive mechanical ventilation calculated in days

8. Remission of respiratory symptoms [ Time Frame: up to 1 month ]\* time to independence from oxygen therapy in days

#### 4 TRIAL DESIGN AND DESCRIPTION

#### 4.1 Trial Design

It is a Multi-Centric, Open label, Two Arm Randomized, Pivotal Phase 2 Trial to Study the Efficacy and Safety of Itolizumab in COVID-19 complications. Patients who have tested positive for virological diagnosis of SARS-CoV2 infection (PCR) are planned to be randomised for enrolment from various centres in India. All eligible patients entering into the study will be randomized in 2:1 ratio to receive the treatment A/B respectively.

#### 4.2 Subject Selection

Patients who have tested positive for virological diagnosis of SARS-CoV2 infection (PCR) are planned to be randomised for enrolment from various centres in India.

#### 4.3 Inclusion Criteria

- 1. Male or female adults above 18 years (not tested in children yet)
- 2. Informed consent for participation in the study
- 3. Confirmed virological diagnosis of SARS-CoV2 infection (RT-PCR)
- 4. Hospitalized due to clinical worsening of COVID-19 infection
- 5. Oxygen saturation at rest in ambient air ≤94%
- 6. Patients who are in moderate to severe ARDS as defined by PaO2/Fio2 ratio of < 200 or more than 25% deterioration from the immediate previous value.
- 7. Baseline serum ferritin level ≥ 400 ng/mL or IL-6 levels greater than 4 times ULN, if known

Note: Either of Inclusion number 6 or 7 is required for inclusion of the patient into the study. Since there is logistical delay in getting results in time, biomarker data as inclusion criteria may be used if already known.

#### 4.4 Exclusion Criteria

- 1. Known severe allergic reactions to monoclonal antibodies
- 2. Active tuberculosis (TB) infection
- 3. History of inadequately treated tuberculosis or latent tuberculosis

Note: Latent tuberculosis should be excluded based on history, physical examination and chest x ray before dosing (day 1). QuantiFERON TB also should be performed, however considering criticality of patient condition, patient can be dosed without QuantiFERON TB test results. If


<sup>\*</sup> Applicable for both arms

QuantiFERON TB test is positive, then continuation of patient in the study is investigator's discretion considering benefit-risk evaluation with the sponsor.

- 4. In the opinion of the investigator, progression to death is highly probable, irrespective of the provision of treatments
- 5. Patient on invasive mechanical ventilator support.
- 6. Have received oral anti-rejection or immune-suppressive drugs within the past 6 months Note: Patient receiving oral anti-rejection or immune-suppressive drugs regularly in the last 6 months will be excluded. Patient will be included if received short course of steroids.
- 7. Participating in other drug clinical trials like using anti-IL-6 therapy like tocilizumab (participation in COVID-19 anti-viral trials may be permitted if approved by Sponsor)
- 8. Patient on treatment of anti-IL-6 or plasma therapy as a part of supportive care
- 9. Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination
- 10. Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
- 11. Patients with known history of Hepatitis B, Hepatitis C or HIV
- 12. Absolute Neutrophils count (ANC) < 1000 / mm<sup>3</sup>
- 13. Platelet count < 50,000 / mm3
- 14. Absolute Lymphocyte count (ALC): <500/mm3

Note: ANC, ALC and platelet counts can be done in local lab in the hospital.

#### 4.5 Sample Size, Treatment Assignment, Randomization

Approximately 30 patients are considered sufficient to explore the study objectives and will be included in this study (number of patients may be increased if there is benefit observed in initial cohort of patients. There is no formal sample size calculation estimated). All eligible patients entering into the study will be randomized in 2:1 ratio to receive the treatment A/B respectively. A computer derived randomization schedule is planned to be generated using appropriate system e.g. SAS to assign patient to treatment groups. Randomization will be central and appropriate system (e.g. remote telephone based, computer-based email, sealed envelope) will be used to distribute randomization schedule to the site Note: If the patient is randomised to Arm A and is not initiated itolizumab or not administer one full infusion, is then not considered randomized. The same randomisation code will be used for the subsequent subject in that particular site.

#### 5 Protocol Deviation

Deviations from the protocol, including deviations of inclusion/exclusion criteria will be assessed as 'major' or 'minor' in agreement with Medical Team. Refer to "Guidance Document for Protocol Deviation Reporting and Specifications" for details. All protocol deviations will be appropriately captured in CSR

### **6** General Aspects for Statistical Methods

In general, metric variables and derived parameters will be presented using descriptive summary statistics including arithmetic mean, standard deviation, median, minimum and maximum.


Categorical variables will be presented using descriptive summary statistics including number of patients and percentages. Percentages of patients will be based on non-missing values. The presentation will be by treatment group. Individual values as well as minimum and maximum will be presented with the same number of decimal places as the raw data. Derived parameter will have as many decimal places as the measured number with the smallest number of decimal places. Descriptive statistics, such as arithmetic/geometric mean and median will be presented with an additional decimal place and standard deviation with two additional decimal places as the raw or derived data. All relevant subject data will be included in the listings; and all subjects entered into the database will be included in subject data listings .SAS 9.4 or any other validated software will be used for analysis purpose and generating Tables, Listings & Figures. P-values less than 0.05 may be reported as statistically significant.

The formatting of the final version of a table, figure, or listing may differ from what is presented in the mock shell or the presentation of the results may be changed, however the key content will remain unchanged. dditional tables, figures, and listings may be generated to supplement the planned output.

#### 7 Analysis Population

ITT/FAS population: Patients randomized (in Arm B) and received at least one full dose of Itolizumab (in Arm A)

Safety population: Patients randomized (in Arm B) and received partial or full dose of Itolizumab (in Arm A)

### 8 Demography other baseline Characterstics

Demographic characteristics including age, gender, race, and ethnicity will be summarized for ITT/FAS populations. Baseline is defined as the last observed value/data before the patient receives study drug for the first time or randomized (in Arm B)

Vital signs such as height, weight, pulse, temperature, respiratory rate, systolic blood pressure, diastolic blood pressure, PaO2/FiO2, FiO2, SpO2, mean arterial pressure & GCS score will be summarized.

Medical history, Physical Examination & concomitant medications will be summarized using counts and percentage. Additionally, prognostic markers and few key laboratory parameters will be summarized.

# 9 Efficacy Evaluation **Primary Efficacy Evaluation**

Proportion of patients with deterioration of lung function as measured by Stable SpO2 without increasing FiO2 and Stable PaO2 without increasing FiO2 will be summarized using count and


percentage. The difference between two proportion with its 95% Confidence interval and

a statistically significant difference between two proportions.

Reduction of endo-tracheal intubation rate, measured as rate of patients needing intubation will be summarize using descriptive statistics.

associated p-values may be presented, if p-value is less than 0.05 it can be concluded that there is

Reduction in proportion of patients who need/ Non-invasive ventilation / Invasive mechanical ventilation/high glow nasal oxygen will be summarized using count & percentage.

One-month mortality rate between the two arms will be summarized. The difference between two rates with its 95% Confidence interval and associated p-values may be presented, if p-value is less than 0.05 it can be concluded that there is a statistically significant difference between two-rates.

Change in inflammatory markers like CRP (C-reactive protein) level, d-Dimer, ferritin etc will be summarize with descriptive statistics. Change from Baseline may be presented along with 95% CI.

#### **Secondary Efficacy Evaluation**

Biomarkers (IL-6, TNF-a, IL1, IL17, etc...) will be summarize using summary statistics.

Lymphocyte count will be summarized using count & percentage.

PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio) calculated from arterial blood gas analyses. Radiological response will be summarized in descriptive manner.

Duration of hospitalization will be summarized using descriptive statistics.

Time to independence from non-invasive mechanical ventilation and from oxygen therapy will be summarize using summary statistics.

Biomarkers (IL-6, TNF-a, IL1, IL17, etc...) Lymphocyte count, CRP (C-reactive protein) level, PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio), will be summarized with descriptive statistics. Change from Baseline will be presented along with 95% CI for the difference between two treatments will be reported.

Radiological response, Duration of hospitalization & Remission of respiratory symptoms will be summarized using descriptive statistics.

Number of participants with treatment-related side effects as assessed by Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 graded according to CTCAE criteria (v5.0) will be summarized based on frequency and proportion of total subjects, by system organ class and preferred term. Proportion of subjects with IRR in both the arm will be presented. An overall summary of deaths will be presented by treatment arms.


## 10 Other Evaluations

#### **Additional Safety Evaluation**

Additional safety analysis will be provided by treatment group, by severity, by outcome and related to study drug. Events will be summarized with descriptive statistics (count & percentage).

#### **Laboratory Evaluations**

For haematology and biochemistry variables, descriptive summaries of observed values and changes from baseline will be presented by treatment arm. Numerical variables will be described by number of subjects, mean, standard deviation, median, minimum and maximum and categorical variables will be described by number and percentage.

#### Vital Signs and Physical examination

Descriptive statistics of each vital signs parameter will be presented for the Safety Population, showing the observed visit and change from baseline to each visit value. These summaries statistics (N, mean, SD, median and Min, Max) will be presented by visit for each treatment arm

#### 11 Interim Study Report

Data will be provided to DSMB (constituted prior to first patient screened) on a periodic basis. Based on DSMB recommendation, interim clinical study report may be prepared and submitted to DCGI/regulatory agencies.

### **12** Key Definitions

For few assessments (weight, physical examination, vital signs haematology, biochemistry Chest X Ray/CT scan), screening assessments will be considered as baseline assessment (as day 1).

#### Stable SpO2:

- Stable SpO2: Defined as absence of increase in FiO2 to maintain Spo2  $\geq$  92%
- Improvement of SpO2: Defined as decrease in FiO2 to maintain SpO2 >92%

#### Stable PaO2:

- Stable PaO2: Defined as up to 10% change in PaO2/FiO2 ratio from baseline
- Improvement of PaO2: Defined as > 10% improvement in PaO2/FiO2 ratio from baseline (including patients weaned off oxygen)

If assessment is missing on particular day then it should be captured from assessment available in next two days.

For lab parameters, if assessment is missing on particular day, then it should be captured from assessment available in  $\pm 2$  days.


# 13 Programming Considerations, Listing of Tables, Figures & Format, Software detail

All tables, data listings, figures (TLFs), and statistical analyses will be generated using SAS® for Windows, Release 9.4 (SAS® Institute Inc., Cary, NC, USA) or any other validated statistical software. One SAS program will be used to create several outputs / a separate SAS program will be created for each output. Output files will be delivered in Word / pdf format.

For few assessments (weight, physical examination, vital signs haematology, biochemistry Chest X Ray/CT scan), screening assessments will be considered as baseline assessment (as day 1).

#### Missing data:

All attempts will be made to collect all data per protocol. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If data points are identified as outliers, sensitivity analyses may be performed to examine the impact of including or excluding the outliers. Subjects who meet fatal outcome during the observing period up to 30 days will be an event. Subjects lost to follow up or withdraw consent during the observing period, will be censored at last assessment. Patient data will be censored at the time of their last observed assessment in case of lost to follow up, withdrawal consent or after 30 days of enrolment.

Following Rules may be applied for the derivation of efficacy endpoints

- Patients who discharged from hospital (with improvement, Off O2), the status at discharge will be carried forward.
- Patients who lost to follow up will be considered as Non evaluable (NE)
- Patients who worsen or met fatal outcome, status at event will be carried forward.

Note: Telephonic improvement of weaning of O2 will be considered as improved.

These rules will be applied to analyse following endpoint:

Proportion of patients with deterioration of lung function as measured by:

- Stable SpO2 without increasing FiO2
- Stable PaO2 without increasing FiO2


#### **Listing of Tables, Figures & Format**

Table, figure, and listing shells are presented in Appendices 14. The formatting of the final version of a table, figure, or listing may differ from what is presented in the shell or the presentation of the results may be changed, however the key content will remain unchanged. Additional summaries/data points may be included in the final version of a table, figure, or listing, as well. Additional tables, figures, and listings may be generated to supplement the planned output.

#### **Software Detail**

SAS version 9.4 or any validated statistical software will be used to generate all tables, figures and listings.

#### 14 Tables and mock shells

#### **14.1.1** Screening Failures

| | Overall |
|--------------------------------------------------------------|-------------|
| | N (%) |
| Total Screened Subjects | XX (XX.X %) |
| Screen Failures | XX (XX.X %) |
| Total Randomized Subject | XX (XX.X %) |
| Subject met Inclusion Criteria or met Exclusion Criteria | XX (XX.X %) |
| Subject not met Inclusion Criteria or met Exclusion Criteria | XX (XX.X %) |
| Others | XX (XX.X %) |
| Withdrawal Informed Consent | XX (XX.X %) |
| Lost to Follow-Up | XX (XX.X %) |

Note: XX patients could not complete first dosing hence replaced as per the protocol.


# **14.1.2** Disposition of Patients

| Disposition | Arm A<br>[n (%)] | Arm B<br>[n (%)] |
|---|---|---|
| Randomized | XX (XX.X %) | XX (XX.X %) |
| ITT/FAS Population | XX (XX.X %) | XX (XX.X %) |
| Safety Population | XX (XX.X %) | XX (XX.X %) |
| Completed the study | XX (XX.X %) | XX (XX.X %) |
| Completed 30 days follow up in hospital | | |
| Early discharged* | | |
| Discontinued | XX (XX.X %) | XX (XX.X %) |
| Reasons for Discontinuation | | |
| Adverse event | XX (XX.X %) | XX (XX.X %) |
| Death | XX (XX.X %) | XX (XX.X %) |
| Physician decision | XX (XX.X %) | XX (XX.X %) |
| As per Protocol | XX (XX.X %) | XX (XX.X %) |
| Lost to follow up | XX (XX.X %) | XX (XX.X %) |
| Subject/Guardian decision | XX (XX.X %) | XX (XX.X %) |
| Diagnosis of COVID 19 by RT-PCR | | |
| Positiive | XX (XX.X %) | XX (XX.X %) |
| Negative | XX (XX.X %) | XX (XX.X %) |
| Not Available | XX (XX.X %) | XX (XX.X %) |

<sup>\*</sup> Patients discharged early due to clinical improvement and government policy during the study.


## 14.1.3 Subject Disposition by Centre

| Center Number | Arm A<br>[n (%)] | Arm B<br>[n (%)] |
|---------------|------------------|------------------|
| 1 | XX (XX.X %) | XX (XX.X %) |
| 2 | XX (XX.X %) | XX (XX.X %) |
| 3 | XX (XX.X %) | XX (XX.X %) |
| 4 | XX (XX.X %) | XX (XX.X %) |

# 14.1.4 Summary of Demographic Characterstics

| | Arm A | Arm B |
|-------------|--------------|--------------|
| | [n (%)] | [n (%)] |
| Age (years) | | |
| N | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| Sex, n (%) | | |
| Male | XX (XX.X %) | XX (XX.X %) |
| Female | XX (XX.X %) | XX (XX.X %) |
| Race, n (%) | | |
| Asian | XX (XX.X %) | XX (XX.X %) |
| Black | XX (XX.X %) | XX (XX.X %) |
| Ethnicity | | |
| Hispanic | XX (XX.X %) | XX (XX.X %) |
| East Asian | XX (XX.X %) | XX (XX.X %) |


## 14.1.5 Summary of Concomitant Medication by treatment group

| | Arm A<br>(N=XX)<br>[n (%)] | Arm B<br>(N=XX)<br>[n (%)] |
|---|---|---|
| Any medication taken | | |
| Yes | XX (XX.X %) | XX (XX.X %) |
| No | XX (XX.X %) | XX (XX.X %) |
| ATC | | |
| XXXXX | XX (XX.X %) | XX (XX.X %) |
| XXXXX | XX (XX.X %) | XX (XX.X %) |
| Medication Name | XX (XX.X %) | XX (XX.X %) |
| XXXXXXXXX | XX (XX.X %) | XX (XX.X %) |
| XXXXXXXXX | XX (XX.X %) | XX (XX.X %) |
| XXXXXXXXX | XX (XX.X %) | XX (XX.X %) |
| XXXXXXXXX | XX (XX.X %) | XX (XX.X %) |
| XXXXXXXXX | XX (XX.X %) | XX (XX.X %) |
| XXXXXXXXX | XX (XX.X %) | XX (XX.X %) |

## 14.1.6 Summary of Medical History

| | Arm A<br>(N=XX)<br>[n (%)] | Arm B<br>(N=XX)<br>[n (%)] |
|---|---|---|
| Diagnosis of COVID 19 by RT-PCR Positive , n (%) | XX (XX.X %) | XX (XX.X %) |
| Duration of COVID-19 related symptoms at enrolment | | |
| N | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| Patients with co-morbidities | | |
| Diabetes Mellitus | XX (XX.X %) | XX (XX.X %) |
| Hypertension | XX (XX.X %) | XX (XX.X %) |
| Others | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |


#### **Summary of Vital Parameters and change from Baseline** 14.1.7

| Variable | Visit | Arm A<br>(N=XX)<br>[n (%)] | Arm B<br>(N=XX)<br>[n (%)] |
|---|---|---|---|
| Weight (kg) | Baseline | | |
| 8 (8) | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | 48 hours | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | Change from Baseline | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |

Note: \*: repeated for Weight, Body Temperature, Pulse, Systolic, Diastolic, Respiratory Rate, PaO2/FiO2, FiO2, SpO2, Mean Arterial Pressure, Glasgow Coma Scale, PaO2 etc

# Repeated for Day 7, Day 14, Day 21, Day 30 and EOS

 Final

# 14.1.8 Summary of Laboratory Test Results and Change from Baseline: Hematology

| Test | Visit | Arm A<br>(N=XX)<br>[n (%)] | Arm B<br>(N=XX)<br>[n (%)] |
|---|---|---|---|
| Haematocrit* % | Baseline <sup>&amp;</sup> | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | Day 7 | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | Change from Baseline&& | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| • | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |

<sup>&</sup>amp;: Repeat for day 14, Day 21, 30/EOS for all applicable parameters,

&&: Repeat for Day 14, Day 21, Day 30/EOS Change from Baseline

# 14.1.9 Summary of Laboratory Test Results and Change from Baseline: Biochemistry


<sup>\*:</sup> Haemoglobin, Total leukocyte count, Platelet count, Absolute lymphocyte count, Absolute neutrophil count, Basophils- Differential, Eosinophils- Differential, Lymphocytes- Differential, Monocytes- Differential and Neutrophils- Differential.etc

SAP Final, Date: 29-JUN-2020

| Variable | Time point | Visit | Arm A<br>(N=XX)<br>[n (%)] | Arm B<br>(N=XX)<br>[n (%)] |
|---|---|---|---|---|
| Blood Urea* | Predose | Baseline <sup>&amp;</sup> | | |
| | | N | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX |
| | | 12-24 hours | | |
| | | N | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX |
| | | Change from Baseline | | |
| | | N | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX |
| | 12-24Hrs Post<br>Dose | Day 7 <sup>&amp;&amp;</sup> | | |
| | | N | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX |

<sup>&</sup>amp;: Repeat for day 14, Day 21, 30/EOS for all applicable parameters , Change from Baseline, Week 3, Change from Baseline, Week 4 and Change from Baseline


<sup>&</sup>amp;&: Repeat for Day 14, Day 21, Day30/EOS 2, Change from Baseline,

<sup>\*:</sup> Serum Bilirubin, AST (SGOT), ALT (SGPT), ALP, Serum Albumin, LDH, HDL, LDL, Triglycerides, Total Cholesterol, Serum creatinine, Procalcitonin, d-Dimer, Trop-I, Ferritin etc.

# 14.1.10 Hospitalization

| | Arm A<br>(N=XX)<br>[n (%)] | Arm B<br>(N=XX)<br>[n (%)] |
|---|---|---|
| Was patient hospitalized during study? | | |
| Yes | XX (XX.X %) | XX (XX.X %) |
| No | XX (XX.X %) | XX (XX.X %) |
| Discharged During study | | |
| Yes | XX (XX.X %) | XX (XX.X %) |
| No | XX (XX.X %) | XX (XX.X %) |
| N/A | XX (XX.X %) | XX (XX.X %) |
| Was patient in Intensive Care Unit during this hospitalization period | | |
| Yes | XX (XX.X %) | XX (XX.X %) |
| No | XX (XX.X %) | XX (XX.X %) |


# 14.1.11 Duration of hospitalization and ICU stay

| | Arm A<br>[n (%)] | Arm B<br>[n (%)] |
|---|---|---|
| No of days of hospitalization | | |
| N | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| No of days of hospitalization during study | ŕ | |
| N | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| No of days of ICU | | |
| N | Xxx | Xxx |
| Mean (SD) | Xxx | Xxx |
| Median | Xxx | Xxx |
| Min, Max | Xxx | Xxx |
| No of days of ICU during study | | |
| N | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| Time to independence from non-invasive mechanical ventilation calculated in days | | |
| N | Xxx | Xxx |
| Mean | Xxx | Xxx |
| Median | Xxx | Xxx |
| Min, Max | Xxx | Xxx |
| Duration in Days for independence from oxygen therapy | | |
| N | Xxx | Xxx |
| Mean | Xxx | Xxx |
| Median | xxx | Xxx |
| Min, Max | xxx | Xxx |


# 14.1.12 Summary of Study Treatment: Itolizumab treatment details in Arm

#### A

| A | |
|--------------------------------------|--------------|
| | Arm A |
| Dose | |
| N | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Min, Max | XX, XX |
| No of infusion received during study | |
| 1 | XX (XX.X %) |
| 2 | XX (XX.X %) |
| 3 | XX (XX.X %) |
| 4 | XX (XX.X %) |
| Infusion interrupted | |
| Yes | XX (XX.X %) |
| No | XX (XX.X %) |
| Reason for interruption | |
| XXXX | XX (XX.X %) |
| XXXX | XX (XX.X %) |
| XXXX | XX (XX.X %) |
| Regimen administered | |
| Weekly | XX (XX.X %) |
| Alternate weekly | XX (XX.X %) |
| Dose deferred | |
| Yes | XX (XX.X %) |
| No | XX (XX.X %) |
| Reason | |
| XXXX | XX (XX.X %) |
| XXXX | XX (XX.X %) |
| XXXX | XX (XX.X %) |


# 14.1.13 Summary of BSC treatment details in both arms

| | Arm A | Arm B |
|-----------------|-------------|-------------|
| | n (%) | n (%) |
| Antibiotics | | |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| Antivirals | | |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| HCQ | XX (XX.X %) | XX (XX.X %) |
| Heparin | XX (XX.X %) | XX (XX.X %) |
| Glucocorticoids | | |
| Supplements | XX (XX.X %) | XX (XX.X %) |
| IV fluids | XX (XX.X %) | XX (XX.X %) |
| Others | | |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |
| XXXX | XX (XX.X %) | XX (XX.X %) |


#### 14.2 Primary outcome measures

## **14.2.1 Primary Outcome Measures**

| Visit* | | Arm A<br>(N=XX) | Arm B (N=XX) |
|---|---|---|---|
| Baseline | patients with Stable SpO2 without increasing FiO2 | XX (XX.X %) | XX (XX.X %) |
| | patients with Stable PaO2 without increasing FiO2 | XX (XX.X %) | XX (XX.X %) |

<sup>\*</sup>day 7, day 14, day 21 and day 30/EOS or all available visits

## 14.2.2 Proportion of patients needed intubation during the study

| | Arm A<br>(N=XX) | Arm B (N=XX) |
|---------------------------------|-----------------|--------------|
| Patients needed intubation n(%) | XX (XX.X %) | XX (XX.X %) |

### 14.2.3 Reduction in proportion of patients who need Non-invasive ventilation

| Visit | | Arm A<br>(N=XX) | Arm B (N=XX) |
|---|---|---|---|
| | Patients on Non-invasive ventilation at baseline | XX | XX |
| Day 7 | N | XX | XX |
| | Stable or improved (shifted to bag and mask, NRBM, FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 14 | N | XX | XX |
| Duj II | Stable or improved (shifted to bag and mask, NRBM, FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 21 | N | XX | XX |
| | Stable or improved (shifted to bag and mask, NRBM, FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 30/EOS | N | XX | XX |
| | Stable or improved (shifted to bag and mask, NRBM, FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |


## 14.2.4 Reduction in proportion of patients who need NRBM

| Visit | | Arm A<br>(N=XX) | Arm B (N=XX) |
|---|---|---|---|
| | Patients on NRBM at baseline | XX | XX |
| | | | <del> </del> |
| Day 7 | N | XX | XX |
| | Stable or improved (shifted to FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 14 | N | XX | XX |
| | Stable or improved (shifted to FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 21 | N | XX | XX |
| | Stable or improved (shifted to FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 30/EOS | N | XX | XX |
| | Stable or improved (shifted to FM, nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |

## 14.2.5 Reduction in proportion of patients who need Face Mask

| Visit | | Arm A<br>(N=XX) | Arm B (N=XX) |
|---|---|---|---|
| | Patients on FM at baseline | XX | XX |
| D 7 | | **** | 7777 |
| Day 7 | N | XX | XX |
| | Stable or improved (shifted to nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 14 | N | XX | XX |
| | Stable or improved (shifted to nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 21 | N | XX | XX |
| | Stable or improved (shifted to nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 30/EOS | N | XX | XX |
| | Stable or improved (shifted to nasal canula or off O2) | XX (XX.X %) | XX (XX.X %) |


## 14.2.6 Reduction in proportion of patients who need High Flow Nasal Oxygen

| Visit | | Arm A<br>(N=XX) | Arm B (N=XX) |
|---|---|---|---|
| | Patients on High flow nasal oxygen at baseline | XX | XX |
| Day 7 | N | XX | XX |
| | Stable or improved (off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 14 | N | XX | XX |
| | Stable or improved (off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 21 | N | XX | XX |
| | Stable or improved (off O2) | XX (XX.X %) | XX (XX.X %) |
| Day 30/EOS | N | XX | XX |
| | Stable or improved (off O2) | XX (XX.X %) | XX (XX.X %) |

### 14.2.7 One-month Mortality Rate

| | Arm A | Arm B |
|--------------------------------|-------------|-------------|
| | [n (%)] | [n (%)] |
| Number of patients died | XX (XX.X %) | XX (XX.X %) |
| 95% CI Difference between Rate | XX (XX | X,XX) |
| p-value | X | |

# 14.2.8 Change in inflammatory markers before and after dosing in Treatment ARM A

| | Before dose | 12-24 hrs after dosing |
|---|---|---|
| Serum ferritin | | |
| First dose (n) | | |
| Mean change | | |
| Second dose (n) | | |
| Mean change | | |
| Third Dose (n) | | |
| Mean change | | |
| Fourth Dose (n) | | |
| Mean change | | |
| Programming Note: Repeat for other inflar | nmatory markers: Serum LDH, Ser | um CRP, Serum d-Dimer etc |
| Repeat Table for first, second, third and for | ourth infusion (dose) of Itolizumab | |


#### 14.2.9 Survival status

| | Arm A<br>(N=XX)<br>[n (%)] | Arm A<br>(N=XX)<br>[n (%)] |
|-----------------|----------------------------|----------------------------|
| Survival Status | XX (XX.X %) | XX (XX.X %) |
| Alive | XX (XX.X %) | XX (XX.X %) |
| Dead | XX (XX.X %) | XX (XX.X %) |
| Unknown | XX (XX.X %) | XX (XX.X %) |

# 14.2.10 Summary of Oxygen and SOFA analysis

| Variable | | Arm A<br>(N=XX) | Arm B<br>(N=XX) |
|---|---|---|---|
| | | [n (%)] | [n (%)] |
| Oxygen requirement (L/min) | Week 1* | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | Week2 | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | Change from Week 1 | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| SOFA score | Week 1* | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | Week2 | | |
| | N | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX |
| | Change from Week 1 | | |
| | N | XX | XX |


| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
|-----------|--------------|--------------|
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |

<sup>\*</sup>Repeated for Day 7, day 14, day 21 and Day 30/EOS

# 14.2.11 Ordinal Scale: No and Proportion of patient reduced by 1 or more points

| | Day 7<br>n (%) | Day 14<br>n (%) | Day 21<br>n (%) | Day 30/EOS<br>n (%) |
|---|---|---|---|---|
| Arm A<br>(n=XX) | | | | |
| Arm B<br>(n=XX) | | | | |

## 14.2.12 Respiratory rate over time

| Sr. No. | Arm A ( | N=xx) | Arm B (N=xx) | |
|------------|-------------|-------------|--------------|-------------|
| | Up to 20 | > 20 | Up to 20 | > 20 |
| Baseline | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| Day 2/3 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| Day 7 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| Day 14 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| Day 21 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| Day 30/EOS | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |


## 14.3 Safety Analysis

## 14.3.1 Summary of Subjects with TEAEs by treatment group

| | | No of events | | No of events |
|---|---|---|---|---|
| | ARM A<br>(N=XX)<br>[n (%)] | | ARM B<br>(N=XX)<br>[n (%)] | |
| Description | | | | |
| At least one TEAE | XX (XX.X %) | XX | XX (XX.X %) | XX |
| At least one related TE AE | XX (XX.X %) | XX | XX (XX.X %) | XX |
| At least one Severe/Grade 3 or above TEAE | XX (XX.X %) | XX | XX (XX.X %) | XX |
| At least one related Severe/Grade 3 or above TE AE | XX (XX.X %) | XX | XX (XX.X %) | XX |
| At least one IRR | XX (XX.X %) | XX | XX (XX.X %) | XX |
| At least one TE SAE | XX (XX.X %) | XX | XX (XX.X %) | XX |
| At least one related TE SAE | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Fatal TEAEs | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Fatal AE related to study drug | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Number of patients with dose temporarily stopped at least once | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Number with dose permanently stopped | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Seriousness criteria | | XX | | XX |
| Death | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Life threatening | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Requires in-patient hospitalization or prolongation of existing hospitalization | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Significant disability | XX (XX.X %) | XX | XX (XX.X %) | XX |
| Congenital anomaly or birth defect Other medically important serious event | XX (XX.X %) | XX | XX (XX.X %) | XX |

Note1: TEAE are defined as any AE which started or deteriorated at or after first dose of study treatment

Note2: Includes related AE.

Note 3: n=number of subjects with AEs. Percentages are based on the number of subjects in safety population (N).


## 14.3.2 Treatment Emergent Adverse Event (TEAE) by SOC and PT

| System Organ Class | Preferred term | ARM A<br>(N=XX)<br>[n (%)] | ARM B<br>(N=XX)<br>[n (%)] |
|---|---|---|---|
| No of Subjects with at least one TEAE | | XX (XX.X %) | XX (XX.X %) |
| Any SOC | | XX (XX.X %) | XX (XX.X %) |
| | PT1 | XX (XX.X %) | XX (XX.X %) |
| | PT2 | XX (XX.X %) | XX (XX.X %) |
| SOC1 | | XX (XX.X %) | XX (XX.X %) |
| | PT1 | XX (XX.X %) | XX (XX.X %) |
| | PT2 | XX (XX.X %) | XX (XX.X %) |
| | PT3 | XX (XX.X %) | XX (XX.X %) |
| | | XX (XX.X %) | XX (XX.X %) |

TEAE are defined as any AE which started or deteriorated at or after first dose of study treatment n=number of subjects with AEs. e=number of events. Percentages are based on the number of subjects in safety population Note: System Organ Class and Preferred Term coded as per MedDRA version XX


## 14.3.3 Treatment Emergent Adverse Event (TEAE) by severity

| | Preferred<br>term | | | ARM A<br>(N=XX)<br>[n (%)] | | | | | ARM B<br>(N=XX)<br>[n (%)] | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| System<br>Organ Class | | Mild | Moderate | | Life<br>threatening | Death | Mild | Moderate | | Life<br>threatening | Death |
| Any SOC | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| SOC1 | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT3 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |

## 14.3.4 Treatment Emergent Adverse Event (TEAE) related to study drug

| | Preferred term | ARM A<br>(N=XX)<br>[n (%)] | | ARM B<br>(N=XX)<br>[n (%)] | |
|---|---|---|---|---|---|
| System Organ Class | | Related | Not related | Related | Not related |
| Any SOC | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| SOC1 | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | PT3 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |

## 14.3.5 Treatment Emergent Adverse Event (TEAE) by Outcome

| | System Organ | Preferred | | | Not recovered/not | Recovered/resolved | | |
|---|---|---|---|---|---|---|---|---|
| ARM | oi. | | Recovered/resolved | Recovering/resolving | | with sequelae | Fatal | Unknown |


| Arm A (N=XX) | Any SOC | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
|---|---|---|---|---|---|---|---|---|
| | | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | SOC1 | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT3 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| Arm B (N=XX) | Any SOC | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | SOC1 | | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT2 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | | PT3 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |

## 15. Supplementary Tables

Table S1: Mean Lymphocyte count

| | Baseline | Day 2/3 | Day 7 | Day 14 | Day 21 | Day 30/EOS |
|-------|----------|---------|-------|--------|--------|------------|
| n | | | | | | |
| Arm A | | | | | | |
| Arm B | | | | | | |

Table S2: Mean PaO2/FiO2 ratio

| | Baseline | Day 2/3 | Day 7 | Day 14 | Day 21 | Day 30/EOS |
|-------|----------|---------|-------|--------|--------|------------|
| n | | | | | | |
| Arm A | | | | | | |
| Arm B | | | | | | |

Table S3: Mean PaO2 / FiO2 ratio in Arm A

| | Before dose | 48 hrs after dose |
|-------------------|-------------|-------------------|
| First dose (n) | | |
| PaO2 / FiO2 ratio | | |
| Mean change | | |
| Second dose (n) | | |
| PaO2 / FiO2 ratio | | |
| Mean change | | |
| Third dose (n) | | |
| PaO2 / FiO2 ratio | | |
| Mean change | | |
| Fourth dose (n) | | |


| PaO2 / FiO2 ratio |
|-------------------|
| Mean change |

#### Table S4: Mean PaO2

| | Baseline | Day 2/3 | Day 7 | Day 14 | Day 21 | Day 30/EOS |
|-------|----------|---------|-------|--------|--------|------------|
| Arm A | | | | | | |
| Arm B | | | | | | |

#### Table S5: Mean FiO2 (%)

| | Baseline | Day 2/3 | Day 7 | Day 14 | Day 21 | Day 30/EOS |
|-------|----------|---------|-------|--------|--------|------------|
| Arm A | | | | | | |
| Arm B | | | | | | |

#### Table S6: Mean SpO2 (%)

| | Baseline | Day 2/3 | Day 7 | Day 14 | Day 21 | Day 30/EOS |
|-------|----------|---------|-------|--------|--------|------------|
| Arm A | | | | | | |
| Arm B | | | | | | |

# 16. Listings

## **Listing 16.1.1 Subjects Inclusion**

| Treatment<br>Group | Subje<br>ct ID | Is the subject eligible for study enrolment based on satisfying all inclusion and exclusion criteria requirement? | IN<br>C 1 | IN<br>C 2 | IN<br>C 3 | IN<br>C 4 | IN<br>C 5 | IN<br>C 6 | IN<br>C 7 |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX | | | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | XXXX | X | X | X | X | X | X | X |
| XXXXX | | | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | XXXX | X | X | X | X | X | X | X |

# **Listing 16.1.2 Subjects Exclusion**

| | | Is the subject<br>eligible for<br>study | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | based on<br>satisfying all<br>inclusion and | | | | | | | | | | | | |
| Treatment<br>Group | Subject | exclusion<br>criteria | EXC 1 | EXC 2 | EXC 3 | EXC 4 | EXC 5 | EXC 6 | EXC 7 | EXC 8 | EXC 9 | EXC<br>10 | EXC 11 | EXC |


SAP Final, Date: 29-JUN-2020

| XXXXXX | XXX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

## Listing 16.1.3 Demographic data

| Treatment Group | Subject<br>ID | Age | Was written informed consent obtained? | Date of Informed<br>Consent | Gender | Date of birth | Is subject of child bearing status | Race | Ethnicity |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XX | XXX | XXX | XXXX | XXXX | XXX | XXX | XXX |
| XXXXXX | XXX | XX | XXX | XXX | XXXX | XXXX | XXX | XXX | XXX |

## **Listing 16.1.4 Medical History**

| Treatment<br>Group | Subject<br>ID | Diagnosis of<br>COVID 19 by RT-<br>PCR | Date | Result | Is there any<br>Medical History to<br>be reported | Serial<br>Number | Medical<br>history term | Start<br>Date | Stop Date | Ongoing |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XX | XXXX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | XX | XXXX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX |

## **Listing 16.1.5 Concomitant Medication**

| Treatment<br>Group | Subject<br>ID | Were any medication(s) taken? | Medication<br>Name | Indication | Start<br>Date | End<br>Date | Ongoing<br>at final<br>exam | Frequency | Route | Dose | Dose<br>units |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX | XX | XXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX | XX | XXX |

# **Listing 16.1.6 Disposition of Subjects**

| Treatment<br>Group | Subject<br>ID | Is the subject<br>eligible to<br>participate in<br>treatment<br>phase? | Did the subject complete study? | If No, primary<br>reason for<br>discontinuation | Date of last contact | Date of consent withdrawn | Diagnosis<br>of COVID<br>19 by RT-<br>PCR | Date | Result |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX |


## **Listing 16.1.7 Vital Parameters**

| Treatm<br>ent<br>Group | Subj<br>ect<br>ID | Date of<br>assessm<br>ent | Time of assessm ent | V<br>isi<br>t | Was<br>assessment<br>performed? | He<br>ig<br>ht | W<br>eig<br>ht | Body<br>Tem<br>pe<br>ratur<br>e | P<br>ul<br>se | Blood<br>Pressu<br>re | Resp<br>irato<br>ry<br>Rate | Pa<br>O<br>2<br>/F<br>iO<br>2 | Fi<br>O<br>2 | S<br>p<br>O<br>2 | M<br>A<br>P | G<br>C<br>S | P<br>a<br>O<br>2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX<br>XX | XX<br>X | XXXX | XX | X<br>X<br>X | XXXX | X<br>X<br>X | X<br>X | XXX | X<br>X<br>X | XXX | XX<br>X | X<br>X.<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X |
| XXXX<br>XX | XX<br>X | XXXX | XX | X<br>X<br>X | XXXX | X<br>X<br>X | X<br>X | XXX | X<br>X<br>X | XXX | XX<br>X | X<br>X.<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X |

## **Listing 16.1.8 Biomarker**

| Treatment<br>Group | Subject<br>ID | Visit | Was blood<br>sample<br>collected pre<br>dose? | Date of sample<br>collected Pre-<br>Dose | Time of sample collected pre dose | Was blood sample collected 12-24 Hours post dose? | Date of sample<br>collected Post-<br>Dose | Time of sample<br>collected 24<br>Hours post dose |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXXX | XXXX | XX | XXX | XXXX | XX |
| XXXXXX | XXX | XXX | XXXX | XXXX | XX | XXX | XXXX | XX |

# **Listing 16.1.9 Haematology**

| Tre<br>atm<br>ent<br>Gro<br>up | Su<br>bj<br>ec<br>t<br>ID | V<br>i<br>s<br>i<br>t | Was<br>blood<br>sample<br>collected<br>pre dose | Date of<br>sample<br>collecte<br>d Pre-<br>Dose | Time of sample collecte d pre dose | Was blood<br>sample<br>collected<br>12 Hours<br>post dose | Date of<br>Sample<br>collecte<br>d Post<br>dose | Time of<br>sample<br>collected<br>12 Hours<br>post | Tes<br>t<br>Par<br>am<br>eter | Res<br>ult-<br>PRE<br>-<br>DO<br>SE | Result<br>-<br>12Hrs<br>POST<br>DOSE | Lowe<br>r<br>Refer<br>ence<br>Rang<br>e | Uppe<br>r<br>Refer<br>ence<br>Rang<br>e | U ni t (S I) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX<br>XX<br>XX | X<br>X<br>X | X<br>X<br>X | XXX | XXXX | XX | XXX | XXXX | XX | XX<br>XX<br>X | XX<br>X | XXX | XXX | XXX | X<br>X |
| XX<br>XX<br>XX | X<br>X<br>X | X<br>X<br>X | XXX | XXXX | XX | XXX | XXXX | XX | XX<br>XX<br>X | XX<br>X | XXX | XXX | XXX | X<br>X |

Note: provide the listing for Haematology parameters as per available data

## **Listing 16.1.10 Biochemistry**

| | | | | | | Was | | Time of | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Was | Date of | | blood | Date of | sample | | | | | | |
| | | | blood | sample | Time of | sample | Sample | collected | | | Result- | | | ł |
| | | | sample | collected | sample | collected | collected | 12 | | Result- | 12Hrs | Lower | Upper | ĺ |
| Treatment | Subject | | collected | Pre- | collected | 12 | Post | Hours | Test | PRE- | POST | Reference | Reference | Unit |
| Group | ID | Visit | pre dose | Dose | pre dose | Hours | dose | post | Parameter | DOSE | DOSE | Range | Range | (SI) |


| | | | | | | post<br>dose | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXXX | XX | XXX | XXXX | XX | XXXXX | XXX | XXX | XXX | XXX | XX |
| XXXXXX | XXX | XXX | XXX | XXXX | XX | XXX | XXXX | XX | XXXXX | XXX | XXX | XXX | XXX | XX |

Note: provide the listing for Haematology parameters as per available data

## **Listing 16.1.11 Study Treatment - Itolizumab**

| Treatment<br>Group | Subject<br>ID | Date<br>of<br>dose | Dose | Frequency | Route | Start<br>Time of<br>infusion | End<br>Time of<br>infusion | Was<br>Infusion<br>interrupted? | Reason for infusion interruption | Stop Time<br>of infusion<br>interruption | Restart<br>Time of<br>infusion | Type<br>of<br>change | Reason<br>for<br>change | Was<br>premedication<br>Hydrocortison<br>administered |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX | XXXX | XXXX | XXXX |

## **Listing 16.1.12 Study Treatment - Supportive Care/Oxygen Therapy**

| Tr ea tm en t Gr ou p | S u b j e c t I D | Na<br>m<br>e<br>of<br>tre<br>at<br>m<br>en<br>t | St art da te of D os e | En d da te of D os e | D<br>o<br>s<br>e | F r e q u e n c y | R o u t e | S t a r t T i m e o f i n f u s i o n | Wa<br>s<br>infu<br>sio<br>n<br>inte<br>rru<br>pte<br>d | Reas<br>on<br>for<br>infus<br>ion<br>inter<br>rupti<br>on | Stop<br>time<br>of<br>infus<br>ion<br>interr<br>uptio<br>n | Res<br>tart<br>Ti<br>me<br>of<br>inf<br>usi<br>on | Deli<br>very<br>mod<br>e for<br>inha<br>latio<br>n | Da<br>te<br>of<br>int<br>ub<br>ati<br>on | Sta<br>rt<br>Ti<br>me<br>of<br>intu<br>bati<br>on | Da<br>te<br>of<br>ex<br>tu<br>ba<br>tio<br>n | Sta<br>rt<br>Ti<br>me<br>of<br>ext<br>uba<br>tion | Was<br>weanin<br>g from<br>mechan<br>ical<br>ventilat<br>ion<br>done? | D<br>at<br>e<br>of<br>w<br>ea<br>ni<br>ng | Ti<br>m<br>e<br>of<br>w<br>ea<br>ni<br>ng | Re<br>as<br>on<br>for<br>ch<br>an<br>ge |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | S | | | | | | | | | |
| X<br>X<br>X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | XX<br>X | XX<br>XX | XXX<br>X | XX<br>XX | XX<br>XX | X<br>X<br>X<br>X | XX<br>XX | X<br>X<br>X<br>X | XX<br>XX | XXXX | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X |
| X<br>X<br>X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | X<br>X<br>X | XX<br>X | XX<br>XX | XXX<br>X | XX<br>XX | XX<br>XX | X<br>X<br>X<br>X | XX<br>XX | X<br>X<br>X<br>X | XX<br>XX | XXXX | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X |


## Listing 16.1.13 Chest X Ray/CT Scan

| Treatment<br>Group | Subject ID | Was CHEST X<br>RAY<br>performed? | Date of assessment | CHEST X<br>RAY | comments | CT SCAN | comments |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | XXX | XXXX | XXX | XXX | XXX | XXX |

## **Listing 16.1.14 Adverse Event (Part1)**

| Treatment<br>Group | Subject<br>ID | Were any<br>adverse<br>events<br>reported? | Adverse<br>event<br>number | Adverse<br>event<br>term | Does this<br>AE meet<br>definition<br>of SAE? | Seriousness<br>criteria | Severity<br>of event<br>as per<br>CTCAE<br>ver 4.03 | Reasonable<br>possibility<br>that AE<br>related to<br>Study Drug | Start<br>Date | End date |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | XXX | XXX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX |

## **Listing 16.1.15 Adverse Event (Part-2)**

| Treatment<br>Group | Subject<br>ID | Is it a<br>study drug<br>infusion<br>site<br>reaction? | Relationship<br>to study drug | If "Unlikely/Unrelated" to study drug, alternative etiology | Action<br>taken on<br>Study<br>Drug | Did this AE lead<br>to<br>discontinuation<br>from the study | Was any concomitant medication taken for this AE? | Outcome |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

## **Listing 16.1.16 Hospitalization**

| | | | | | | Was patient in | | | If yes, | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Intensive Care | | | number | | |
| | | Was patient | | | | Unit during | | Date of | of days | | |
| | | hospitalized | | | Ongoing at | this | Date of | discharge | in | Primary | Were these |
| Treatment | Subject | during | Date of | Date of | final | hospitalization | admission | from | Intensive | reason for | additional organ |
| Group | ID | study? | Admission | Discharge | examination | period | to ICU | ICU | care unit | hospitalization | support needed? |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX |


#### **Listing 16.1.17 Survival Status**

| Treatment Group | Subject ID | Date of assessment | Survival Status | Last known date subject alive | If Subject died,<br>kindly record-<br>Date of Death | Time of death |
|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX |

### **Listing 16.1.18 SOFA Score**

| Treatment<br>Group | Subject<br>ID | Respiratory<br>system<br>(PaO2/FiO2) | Central<br>Nervous<br>system<br>(Glasgow<br>Coma Scale) | Cardiovascular system<br>(Mean arterial pressure<br>(MAP) OR<br>administration of<br>vasopressors required) | Liver<br>(Bilirubin<br>(mg/dl)<br>[µmol/L]) | Coagulation<br>(Platelets ×103/ml) | Kidney<br>(Creatinine<br>(mg/dl)<br>[µmol/L]; urine<br>output) |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

## **Listing 16.1.19 Ordinal Scale**

| Treatment Group | Subject ID | Patient state | Descriptor | Score |
|-----------------|------------|---------------|------------|-------|
| XXXXXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | XXX | XXX | XXX |

## Graphs

• Figure 1: Disposition by centres: Bar Graph

• Figure 2: PaO2/FiO2 ratio: Line Graph

• Figure 3: change from baseline for Key Lab parameters: Ferrtin, d-dimer, LDH, CRP, Lymphocyte counts

• Figure 4: KM Curve for time to event endpoints
